CLINICAL TRIAL: NCT01257139
Title: Trial Involving Subjects Over 70 Years of Age With Non Small-cell Lung Cancer of Stage IV and Comparing a "Classical" Strategy of Treatment Allocation, With an"Optimized" Strategy Allocating the Same Treatments
Acronym: ESOGIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EudraCT 2008-008372-13
Record Dates: First submitted 2010-01-21; First posted 2010-12-09 (Estimated); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Non Small-cell Lung Cancer
Keywords: To evaluate a geriatric scale designed to help with treatment; allocation to dual-agent therapy based on platinum or to; single-agent chemotherapy in elderly subjects with advancedstage; NSCLC, based on the time to failure in the two arms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

ARMS (2):
- dual-agent therapy or docetaxel alone (No Intervention): dual-agent therapy based on Carboplatin (Carboplatin-Pemetrexed for non epidermoid forms, Carboplatin-Gemcitabin for epidermoid forms) or Docetaxel alone, according to PS or age
- dual-agent therapy or docetaxel or best supportive care (Experimental): dual-agent therapy based on Carboplatin (Carboplatin-Pemetrexed for non epidermoid forms, Carboplatin-Gemcitabin for epidermoid forms) or Docetaxel alone, or best supportive care, allocated on the basis of a simplified geriatric scale, plus a more thorough geriatric evaluation if necessary
  Interventions: Procedure: Dual-agent therapy or docetaxel alone or best supportive care

INTERVENTIONS:
Procedure: Dual-agent therapy or docetaxel alone or best supportive care — ARM B: (245 patients)
  Treatment if the SGS screening test is negative:
  * non epidermoid tumor:
  * Carboplatin ® AUC 5 on D1 and Alimta ®(pemetrexed) 500 mg/m² D1, D1=D21 with vitamin B9 and B12 supplementation. Maximum of four 3-week cycles.
  * epidermoid tumor:
  * Carboplatin AUC 5 on D1 and Gemcitabin 1000 mg/m² on D1 and D8, D1=D21. Treatment if SGS screening test is positive (cf.table 1): Vulnerable subjects will receive: Taxotere ® (Docetaxel) 38 mg/m² on D1 and D8, D1=D21. Maximum of four 3-week cycles Fragile subjects are patients considered to be at a high risk of complications during chemotherapy; they will therefore receive best supportive care (BSC) with appropriate geriatric management.
  Arms: dual-agent therapy or docetaxel or best supportive care

SUMMARY:
This is a phase III randomized multicenter study involving subjects over 70 years of age with non small-cell lung cancer of IV and a PS of 0, 1 or 2, who have not previously received chemotherapy. The aim is to validate the use of a simplified geriatric scale (SGS) as a screening tool. If the SGS results are normal, the patient will be treated with dual-agent therapy based on platinum (carboplatin + pemetrexed if the histology is non epidermoid, carboplatin + gemcitabin if the histology is epidermoid), with no further geriatric assessment. When the SGS reveals abnormalities, a comprehensive geriatric evaluation (CGE) will be used to define two subpopulations on Balducci's fragility scale, who will receive either monotherapy (docetaxel) or best supportive care.

The strategy based on the SGS will be compared with a treatment algorithm based on standard criteria (PS and age), with no specific geriatric assessment. The main endpoint is the time to treatment failure. The SGS is composed of the Charlson co-morbidity scale, functional assessment based on PS, Katz' ADL scale, Lawton's simplified IADL scale, simplified cognitive assessment with the mini-MMSE according to Schultz-Larsen, a geriatric depression scale (GDS 5), and screening for a geriatric syndrome defined by the existence of dementia, repeated falls, and urinary and fecal incontinence. The SGS will be validated by comparison with the CGE, that will be administered systematically at enrollment. All the SGS items are included in the CGE.

Secondary endpoints will be quality of life (measured with the LCSS and EuroQoL questionnaires), overall survival, the objective response rate, and toxicity. The investigators will also study the predictive power of nutritional indices such as the PINI and the Buzby score with respect to survival, the treatment response, and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically proven NSCLC(adenocarcinoma, epidermoid carcinoma, large-cell carcinoma) of stage IV with histologically or cytologically proven pleurisy or neoplastic pericarditis.
* No previous systemic chemotherapy for lung cancer.
* Presence of at least one measurable target lesion (RECIST rules) in a non irradiated region.
* Age strictly at least 70 years.
* PS 0, 1 or 2.
* Life expectancy sup 12 weeks.
* Creatinine clearance at least 45 ml per min with MDRD Formula (Modification in the Diet in Renal Disease).
* Normal hematologic function: absolute polymorphonuclear neutrophil count > 1.5 . 109 per l and or platelets sup 100 . 109/l, hemoglobin sup 9.5 g per dl
* Normal hepatic function: bilirubin inf 1.5 x normal, SGOT and SGPT inf 2.5 . normal.
* Patients with metastatic relapse (cytologically or histologically proven) of primary lung cancer in a non irradiated region, after surgical excision or local external radiotherapy.
* Prior irradiation is authorized if it involved less than 25 percent of the total bone marrow volume.
* Men must be surgically sterile or must accept the use of an effective contraceptive methodall along and until 6 months after the treatment period
* Signed written informed consent.

Exclusion Criteria:

* Other severe concurrent disorders that occurred during the prior six months before enrollment (myocardial infection, severe or unstable angor, coronarian or peripheric arterial bypass operation, NYHA class 3 or 4 congestive heart failure, transient or constituted cerebral ischemic attack, at least grade 2 peripheral neuropathy, stomach ulcer, erosive oesophagitis or gastritis, psychiatric or neurological disorders preventing the patient from understanding the trial, uncontrolled infections).
* Another previous or concomitant cancer, except for basocellular cancer of the skin or treated cervical cancer in situ, or appropriately treated localized lowgrade prostate cancer (Gleason score inf 6), unless the initial tumor was diagnosed and definitively treated more than 5 years previously, with no evidence of relapse.
* Bronchoalveolar or neuroendocrine or composite cancers
* Superior caval syndrome.
* Presence of symptomatic brain metastases.
* Peripheral neuropathies (grade sup 2).
* Performance status sup 2 (ECOG).
* A significant third liquid part (for example ascitis or pleural effusion) hat can't be controlled with drainage or other procedures before enrollment
* Impossibility to stop a treatment by aspirin (if the dose is more than 1.3 mg per day) or NSAI during 5 days (8 days for molecules with long period action like piroxicam
* Concurrent participation in another clinical trial.
* Definitive contraindication to steroids or folic acid and vitamin B12 if histology is non-epidermoid.
* All concurrent radiotherapy, except for local palliative bone radiotherapy.
* Concurrent administration of one or several other antitumor therapies. Recent vaccination for yellow fever (during the 30 days before enrollment)
* Psychological, familial, social or geographic difficulties preventing follow-up as defined by the protocol.
* Administrative or legal detention.
* Contraindication to the study drugs.
* Concurrent participation in another clinical trial

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 490 (Actual)
Dates: Start 2010-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Time to failure Defined from the date of inclusion to the date of documented progression Or death of any cause Or trial exit for toxicity considered unacceptable by the patient or by the investigator Or withdrawal of consent | date of documented progression up to 6 months

CONTACTS AND LOCATIONS:
Locations (45):
- France (45):
  - CH du Pays d'Aix, Aix-en-Provence
  - CHU Amien Picardie, Amiens
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Centre Hospitalier d'Annecy, Annecy
  - Centre Hospitalier Général de la Fontonne Antibes, Antibes
  - CH de Bastia, Bastia
  - Centre Hospitalier de Beauvais, Beauvais
  - CHU Bordeaux Hôpital Haut Lévêque, Bordeaux Pessac
  - Centre Hospitalier Universaitaire de Brest, Brest
  - HIA Tonnerre, Brest
  - Centre François Baclesse, Caen
  - CH René Dubos - Pontoise, Cergy-Pontoise
  - Centre Hospitalier Charleville mézières, Charleville-Mézières
  - CHI Créteil, Créteil
  - Centre hospitalier de Draguignan, Draguignan
  - Centre Hospitalier de Elbeuf, Elbeuf
  - CH Gap, Gap
  - CH La Roche sur Yon, La Roche-sur-Yon
  - Hôpital A Mignot Le Chesnay, Le Chesnay
  - Centre Omar Lambret, Lille
  - Hôpital du Cluzeau, Limoges
  - CHR Longjumeau, Longjumeau
  - Centre Hospitalier de Bretagne Sud, Lorient
  - Hôpital de la Croix Rousse, Lyon
  - Centre Hospitalier, Mantes-la-Jolie
  - Hôpital Sainte Marguerite, Marseille
  - Institut Paoli-Calmette, Marseille
  - Centre Hospitalier, Martigues
  - Hôpital Saint Farron, Meaux
  - Centre Hospitalier de Mulhouse, Mulhouse
  - CHR Orléans, Orléans
  - Paris Hôpital saint Antoine, Paris
  - Centre Catalan, Perpignan
  - Centre Hospitalier de Périgueux, Périgueux
  - Rennes Hospital University, Rennes
  - CHU Rouen Hôpital Boisguillaume, Rouen
  - Hôpital Charles Nicolle, Rouen
  - Hôpital Yves Le Foll, Saint-Brieuc
  - CHU Saint Etienne - Hôpital Nord, Saint-Etienne
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Centre Hospitalier Général Salon de Provence, Salon-de-Provence
  - Hôpital Font-Pre, Toulon
  - Hôpital d'Instruction des Armées, Toulon Naval
  - CHU Touloues, Toulouse
  - Centre Hospitalier De Villefranche sur Saone, Villefranche-sur-Saône

REFERENCES:
- [Result] Corre R, Greillier L, Le Caer H, Audigier-Valette C, Baize N, Berard H, Falchero L, Monnet I, Dansin E, Vergnenegre A, Marcq M, Decroisette C, Auliac JB, Bota S, Lamy R, Massuti B, Dujon C, Perol M, Daures JP, Descourt R, Lena H, Plassot C, Chouaid C. Use of a Comprehensive Geriatric Assessment for the Management of Elderly Patients With Advanced Non-Small-Cell Lung Cancer: The Phase III Randomized ESOGIA-GFPC-GECP 08-02 Study. J Clin Oncol. 2016 May 1;34(13):1476-83. doi: 10.1200/JCO.2015.63.5839. Epub 2016 Feb 16. PMID 26884557